CLINICAL TRIAL: NCT07280780
Title: Continuous Glucose Monitoring-Based Evaluation of Glycemic Fluctuations Following Epidural Steroid Injections: A Comparative Study by Diabetic Status
Brief Title: CGM-Based Glycemic Analysis After ESI
Acronym: CGMSteroid
Status: Not yet recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: The Korean Pain Society (Unknown)
Responsible Party: Principal Investigator, Sunmin Kim, Clinical Assistant Professor, Korea University Anam Hospital
Other Study IDs: K2025-2728-002
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes (T2DM); Hyperglycemia; Radicular Pain; Spinal Stenosis; Intervertebral Disc Herniation
Keywords: epidural steroid injection; Continuous Glucose Monitoring; Dexamethasone; Glycemic Variability; Time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Spinal Stenosis; Intervertebral Disc Displacement | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D (Type 2 Diabetes): Patients diagnosed with Type 2 Diabetes Mellitus who are scheduled for an epidural steroid injection.
  Interventions: Procedure: Epidural Steroid Injection; Device: Continuous Glucose Monitoring
- Group C (Non-Diabetes): Patients without diabetes who are scheduled for an epidural steroid injection.
  Interventions: Procedure: Epidural Steroid Injection; Device: Continuous Glucose Monitoring

INTERVENTIONS:
Procedure: Epidural Steroid Injection — Administration of 5 mg Dexamethasone via epidural route (cervical or lumbar) under fluoroscopic guidance.
Device: Continuous Glucose Monitoring — A sensor attached to the upper arm to monitor interstitial glucose levels continuously for 15 days.

SUMMARY:
The goal of this clinical study is to learn how blood glucose levels change after an epidural steroid injection (ESI) with dexamethasone in adults. It will specifically compare the glycemic response between patients with type 2 diabetes and those without diabetes.

The main questions it aims to answer are:

Does the injection cause higher or longer-lasting blood glucose elevation in diabetic patients compared to non-diabetic patients? How do the mean glucose level and Time in Range (TIR) change after the injection in both groups?

Researchers will compare a Type 2 Diabetes group to a Non-Diabetes group to see the differences in glycemic fluctuations using a continuous glucose monitoring (CGM) device.

Participants will:

* Wear a small CGM sensor on their arm for about 15 days to monitor blood glucose levels continuously
* Receive an epidural steroid injection containing 5 mg of dexamethasone on Day 3
* Visit the clinic 3 times (Day 1, Day 3, and Day 15) for sensor attachment, the injection procedure, and data collection

DETAILED DESCRIPTION:
Epidural steroid injections (ESIs) are a widely used non-surgical treatment for radicular pain caused by spinal conditions such as herniated discs and spinal stenosis. While effective for pain relief, the systemic absorption of corticosteroids (e.g., dexamethasone) can induce temporary hyperglycemia, which poses potential risks, particularly for patients with type 2 diabetes mellitus (T2DM).

Previous studies on post-ESI hyperglycemia have largely relied on self-monitoring of blood glucose (SMBG), which captures only intermittent glucose data and may miss significant glycemic excursions, such as postprandial spikes or nocturnal hypoglycemia. This study aims to overcome these limitations by using a Continuous Glucose Monitoring (CGM) system to provide a comprehensive, time-series analysis of glycemic fluctuations.

Objectives:

To compare glycemic changes (mean glucose, Time in Range [TIR], Time Above Range [TAR]) following an epidural steroid injection with 5 mg of dexamethasone between a type 2 diabetes group and a non-diabetes control group.

To investigate the correlation between baseline HbA1c levels and the magnitude of post-injection glycemic variability.

Study Design: This is a prospective, observational, comparative study conducted at a single center (Korea University Anam Hospital). A total of 36 participants (18 in the T2DM group and 18 in the Non-DM group) will be enrolled.

Study Procedures:

Visit 1 (Day 1 - Screening & Baseline):

* Participants provide informed consent and undergo screening.
* Baseline HbA1c is measured.
* A CGM sensor (Abbott FreeStyle Libre 2) is attached to the participant's upper arm.
* Participants receive education on CGM use and are instructed to maintain their usual diet and medication.
* Baseline Data Collection: Glucose levels are monitored for 2 days (Day 1-2) to establish a baseline profile before the injection.

Visit 2 (Day 3 - Intervention):

* Participants undergo the scheduled epidural steroid injection (cervical or lumbar) using 5 mg of dexamethasone.
* The procedure is performed under fluoroscopic guidance according to standard clinical practice.

Visit 3 (Day 15 - Follow-up & Data Collection):

* Participants return to the clinic for follow-up.
* The CGM sensor is removed, and the stored glycemic data is downloaded.
* Pain intensity (Numeric Rating Scale, NRS) and any adverse events are recorded.

Statistical Analysis: The primary endpoints (changes in mean daily glucose and TIR) will be analyzed using a Linear Mixed Model (LMM) to account for repeated measures. Fixed effects will include Group (DM vs. Non-DM), Time (Baseline vs. Post-injection), and the Group-by-Time interaction. Patient demographics (e.g., age, BMI) will be included as covariates if significant differences are observed at baseline. A p-value of <0.05 will be considered statistically significant.

This study will provide high-resolution data on the duration and severity of steroid-induced hyperglycemia, contributing to safer pain management protocols for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 60 years.
* Patients scheduled for cervical or lumbar epidural steroid injection at the pain clinic.
* Patients capable of understanding and using a Continuous Glucose Monitoring (CGM) device.

Exclusion Criteria:

* Patients currently taking or administering steroid medications.
* Patients with Type 1 Diabetes Mellitus.
* Patients with Cushing's disease.
* Patients who have received an epidural steroid injection within the last 3 months.
* Patients with a known allergy to contrast media.
* Patients taking anticoagulants or antiplatelet agents.
* Patients unable to use a Continuous Glucose Monitoring (CGM) device.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients visiting the Pain Clinic at Korea University Anam Hospital who are scheduled for cervical or lumbar epidural steroid injections due to spinal pain.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2026-12-17 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Mean Glucose | Baseline (Day 1-2) and up to 12 days post-injection (Day 15)
  The difference in daily mean glucose levels (mg/dL) measured by CGM between the baseline period (Day 1-2) and the post-injection period (Day 3-15).
Change in Time in Range (TIR) | Baseline (Day 1-2) and up to 12 days post-injection (Day 15)
  The difference in the percentage of time (%) spent within the target glucose range (70-180 mg/dL) between the baseline period and the post-injection period.

SECONDARY OUTCOMES:
Change in Numeric Rating Scale (NRS) | Baseline (Day 1) and Day 15
  The change in pain intensity scores reported by participants. The scale ranges from 0 (no pain) to 10 (worst possible pain).
Frequency of Glucose Spikes | Up to 12 days post-injection (Day 15)
  The number of hyperglycemic events defined as glucose levels >180 mg/dL lasting for at least 30 minutes.
Incidence of Nocturnal Hypoglycemia | Up to 12 days post-injection (Day 15)
  The percentage of participants experiencing glucose levels <70 mg/dL during the nighttime period (22:00 to 06:00).
Glucose Variability (Coefficient of Variation) | Up to 12 days post-injection (Day 15)
  The coefficient of variation (%CV) of glucose levels, calculated as the standard deviation divided by the mean glucose, to assess glycemic variability.

CONTACTS AND LOCATIONS:
Overall Officials: Sunmin Kim, M.D., Study Director — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No